CLINICAL TRIAL: NCT06300008
Title: Efficacy of Cetylated Fatty Acid for Alleviating Postoperative Pain After Total Knee Arthroplasty: A Randomized Placebo-controlled Trial
Brief Title: Cetylated Fatty Acid for Reducing Pain After TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, Principle investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OrthoTU13
Record Dates: First submitted 2022-11-24; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain; Postoperative Inflammation
Keywords: Cetylated fatty acid; TKA; Postoperative pain; Inflammation
MeSH Terms: conditions — Pain, Postoperative; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cetylated fatty acid (Experimental): Topical cetylated fatty acid, apply 2 times/day for 6 weeks after operation
  Interventions: Drug: cetylated fatty acid
- Placebo (Placebo Comparator): Topical placebo, apply 2 times/day for 6 weeks after operation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cetylated fatty acid — use approximately 3 cm long of cream per each side of knee, then apply on the operated knee until completely absorb
  Other Names: Cetilar
  Arms: cetylated fatty acid
Drug: Placebo — use approximately 3 cm long of cream per each side of knee, then apply on the operated knee until completely absorb
  Arms: Placebo

SUMMARY:
To compare efficacy of cetylated fatty acid with placebo for reducing postoperative pain after unilateral TKA. The hypothesis is topical cetylated fatty acid can mitigate postoperative pain after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80 years
* Osteoarthritic knee patients underwent unilateral primary TKA
* Participants understand and consent to the protocol of the trial

Exclusion Criteria:

* Inflammatory knee arthritis
* Previous knee surgery or trauma
* Previous knee infection
* Skin problem around the knee such as eczema, psoriasis, wound infection
* Allergy to studied drug

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | post-op Day2
  VAS (0-100) at rest and on motion
Visual analog scale | post-op week2
  VAS (0-100) at rest and on motion
Visual analog scale | post-op week6
  VAS (0-100) at rest and on motion
Visual analog scale | post-op week12
  VAS (0-100) at rest and on motion
inflammatory marker | post-op day2
  ESR and CRP
inflammatory marker | post-op week2
  ESR and CRP
inflammatory marker | post-op week6
  ESR and CRP
inflammatory marker | post-op week12
  ESR and CRP
Knee skin temperature | post-op Day2
  evaluated by digital infrared thermometer at 4 different locations on the anterior aspect of the knee independently (superomedial, superolateral, inferomedial, inferolateral borders of the patella) compared with the contralateral knee
Knee skin temperature | post-op week2
  evaluated by digital infrared thermometer at 4 different locations on the anterior aspect of the knee independently (superomedial, superolateral, inferomedial, inferolateral borders of the patella) compared with the contralateral knee
Knee skin temperature | post-op week6
  evaluated by digital infrared thermometer at 4 different locations on the anterior aspect of the knee independently (superomedial, superolateral, inferomedial, inferolateral borders of the patella) compared with the contralateral knee
Knee skin temperature | post-op week12
  evaluated by digital infrared thermometer at 4 different locations on the anterior aspect of the knee independently (superomedial, superolateral, inferomedial, inferolateral borders of the patella) compared with the contralateral knee

SECONDARY OUTCOMES:
Knee circumference (cm) | post-op Day2
  Measured by tape at midpoint of patella
Knee circumference (cm) | post-op week2
  Measured by tape at midpoint of patella
Knee circumference (cm) | post-op week6
  Measured by tape at midpoint of patella
Knee circumference (cm) | post-op week12
  Measured by tape at midpoint of patella
Knee Range of Motion | post-op Day2
  Flexion and extension angle
Knee Range of Motion | post-op week2
  Flexion and extension angle
Knee Range of Motion | post-op week6
  Flexion and extension angle
Knee Range of Motion | post-op week12
  Flexion and extension angle
Modified WOMAC | post-op week2
  Total & Subscore
Modified WOMAC | post-op week6
  Total & Subscore
Modified WOMAC | post-op week12
  Total & Subscore
Thai forgotten joint score | post-op week2
Thai forgotten joint score | post-op week6
Thai forgotten joint score | post-op week12

CONTACTS AND LOCATIONS:
Overall Officials: Supakit Kanitnate, MD, Principal Investigator — Thammasat University Hospital
Locations (1):
- department of orthopaedic surgery, Faculty of medicine, Thammasat university, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No